CLINICAL TRIAL: NCT03849716
Title: Evaluation of Biomarkers of Atopic Dermatitis in Pediatric Patients Whose Disease is Not Adequately Controlled With Topical Prescription Therapies or When Those Therapies Are Not Medically Advisable
Brief Title: Evaluation of Biomarkers of Atopic Dermatitis in Pediatric Patients (PEDISTAD BIOMARKER STUDY)
Status: Active, not recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: LPS15496; U1111-1207-8876 (Registry Identifier: ICTRP)
Record Dates: First submitted 2019-01-17; First posted 2019-02-21 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Dermatitis Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with atopic dermatitis (AD): Participants included in observational study OBS15333 (atopic dermatitis pediatric registry) who consent to enter this companion study LPS15496. Participants receive AD therapy as part of their usual care as determined by their physician independent of decision to enter either protocol, and neither protocol OBS15333 nor LPS15496 specifies assignment of any drug intervention
  Interventions: Other: Blood sample; Other: Cheek swab

INTERVENTIONS:
Other: Blood sample — Blood samples obtained for biomarker analyses
Other: Cheek swab — Cheek swab obtained for genetic analysis

SUMMARY:
Primary Objective:

To explore associations between biomarkers of atopic dermatitis (AD) and:

* Disease state and time course of AD,
* Disease state and evolution of selected atopic comorbid conditions,
* Effectiveness of specific AD treatments.

DETAILED DESCRIPTION:
The estimated enrollment duration is approximately 2 years, while duration of observation is approximately 5 years.

ELIGIBILITY:
Inclusion criteria:

* Participation in the OBS15333 pediatric atopic dermatitis (AD) registry.
* Signed informed consent by the parent/legally acceptable representative and assent by the participant appropriate to the participant's age.

Exclusion criteria:

Not applicable.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 0 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients with moderate to severe AD whose disease is not adequately controlled with topical therapies or when those therapies are not medically advisable, who are included in observational study OBS15333 and consent to enter this companion study LPS15496.
Sampling Method: Non-Probability Sample
Enrollment: 266 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Biomarker identification: Demographics | Baseline
  Identification of biomarkers associated with demographic characteristics
Biomarker identification: Baseline disease characteristics | Baseline
  Identification of biomarkers associated with disease characteristics at study entry (eg, disease severity, presence of other co-morbidities)
Biomarker identification: Changes in disease severity | Up to 5 years
  Identification of biomarkers associated with disease severity increases/decreases (including remission) over time
Biomarker evaluation: High versus low disease severity across participants | Up to 5 years
  Examination of biomarker expression in participants with high disease severity versus those with low disease severity
Biomarker identification: New presentation or resolution of atopic comorbidity | Up to 5 years
  Identification of biomarkers associated with onset of a new atopic comorbidity or resolution of an existing atopic comorbidity
Biomarker identification: Introduction of new systemic treatment | Up to 5 years
  Identification of biomarkers associated with introduction of new systemic treatment
Biomarker identification: Response to systemic treatment | Up to 5 years
  Identification of biomarkers associated with response to systemic treatment
Biomarker identification: Loss of response to systemic treatment | Up to 5 years
  Identification of biomarkers associated with loss of response to systemic treatment
Biomarker evaluation: Start of systemic therapy early in life versus later in life | Up to 5 years
  Examination of whether biomarker expression in participants who started systemic therapy for AD early in life (within 6 months) differs from those who started it later in life

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (48):
- United States (22):
  - C Squared Research Center Site Number : 8400068, Birmingham, Alabama
  - Cahaba Dermatology Site Number : 8400046, Birmingham, Alabama
  - C2 Research Center, LLC Site Number : 8400071, Montgomery, Alabama
  - Axis Clinical Trials Site Number : 8400025, Los Angeles, California
  - Madera Family Medical Group Site Number : 8400054, Madera, California
  - Fomat Medical Research, Inc. Site Number : 8400033, Oxnard, California
  - Amedica Research Institute, Inc. Site Number : 8400067, Hialeah, Florida
  - Eastern Research, Inc. Site Number : 8400032, Hialeah, Florida
  - Vista Health Research, LLC Site Number : 8400034, Miami, Florida
  - Pediatric & Adult Research Center Site Number : 8400040, Orlando, Florida
  - Georgia Pollens Clinical Research Centers, Inc. Site Number : 8400057, Albany, Georgia
  - IACT Health Site Number : 8400056, Columbus, Georgia
  - Northwestern University Feinberg School of Medicine Site Number : 8400001, Chicago, Illinois
  - NorthShore University HealthSystem Site Number : 8400064, Skokie, Illinois
  - Philip Fried, M.D., PLLC Site Number : 8400029, The Bronx, New York
  - Tiga Pediatrics, PC Site Number : 8400037, The Bronx, New York
  - Cincinnati Children's Hospital Medical Center Site Number : 8400017, Cincinnati, Ohio
  - Dermatology Associates of Mid-Ohio Site Number : 8400052, Marion, Ohio
  - MUSC Site Number : 8400013, Charleston, South Carolina
  - Allergic Disease and Asthma Research Center, PA Site Number : 8400048, Greenville, South Carolina
  - Amarillo Center for Clinical Research Site Number : 8400055, Amarillo, Texas
  - Heights Dermatology and Aesthetic Center Site Number : 8400065, Houston, Texas
- Argentina (5):
  - Investigational Site Number : 0320002, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Investigational Site Number : 0320006, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Investigational Site Number : 0320004, Rosario, Santa Fe Province
  - Investigational Site Number : 0320003, Buenos Aires
  - Investigational Site Number : 0320001, Ciudad Autonoma Bs As
- Australia (2):
  - Investigational Site Number : 0360001, Westmead, New South Wales
  - Investigational Site Number : 0360003, Melbourne, Victoria
- Brazil (6):
  - Universidade Federal do Paraná Site Number : 0760003, Curitiba, Paraná
  - HC - UFPR - Hospital de Clínicas da Universidade Federal do Paraná Site Number : 0760004, Curitiba, Paraná
  - HC - UFPR - Hospital de Clínicas da Universidade Federal do Paraná Site Number : 0760005, Curitiba, Paraná
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre Site Number : 0760002, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Paulo Site Number : 0760006, SÃ£o Paulo, São Paulo
  - Clínica de Alergia Martti Antila Site Number : 0760001, Sorocaba
- Canada (4):
  - Investigational Site Number : 1240007, Calgary, Alberta
  - Investigational Site Number : 1240005, Winnipeg, Manitoba
  - Investigational Site Number : 1240008, Toronto, Ontario
  - Investigational Site Number : 1240006, Montreal, Quebec
- Colombia (2):
  - Investigational Site Number : 1700001, Bogotá
  - Investigational Site Number : 1700004, Bogotá
- France (2):
  - Investigational Site Number : 2500006, Marseille
  - Investigational Site Number : 2500003, Paris
- Mexico (3):
  - Investigational Site Number : 4840003, Monterrey, Nuevo León
  - Investigational Site Number : 4840006, México
  - Investigational Site Number : 4840005, Tlalnepantla
- Netherlands (2):
  - Investigational Site Number : 5280005, Groningen
  - Investigational Site Number : 5280003, Utrecht

IPD SHARING:
Plan to Share IPD: No